CLINICAL TRIAL: NCT01911962
Title: A Prospective Randomized Controlled Study of Natural Orifice Medium-low Rectal Endometriosis Resection
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Wang Shaochuan, Postgraduate, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: nova-0425
Record Dates: First submitted 2013-07-23; First posted 2013-07-30 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Colon Rectal Resection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- transabdominal laparoscope surgery: transabdominal laparoscope surgery
- transvaginal laparoscopic surgery: transvaginal laparoscopic surgery
  Interventions: Procedure: transvaginal laparoscopic surgery

INTERVENTIONS:
Procedure: transvaginal laparoscopic surgery
  Groups: transvaginal laparoscopic surgery

SUMMARY:
To evaluate the postoperative outcome of low medium-low rectal endometriosis: Natural orifice surgery VS transabdominal surgery.

DETAILED DESCRIPTION:
To evaluate the postoperative outcome of low medium-low rectal endometriosis: Natural orifice surgery VS transabdominal surgery.Both of the two kinds of surgery is conventional,but the comparison is still unclear.The investigators divide the patients into two groups, and compare the differences of postoperative outcomes by statistics.

ELIGIBILITY:
Inclusion Criteria:

Childbearing age women,

older than 18 years,

diagnosed with intestinal endometriosis,

rectum clinical symptoms for invalid medical treatment,

dysmenorrhea, dyspareunia dyschezia, infertility, defecate carries blood,

endometriosis in the lower rectum by intraoperative judgment

Exclusion Criteria:

without endometriosis rectum,

history of colorectal surgery,

intolerance to laparoscopic surgery

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Inpatients
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2011-01; Primary Completion 2012-02 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
rectovaginal fistula | one year
  number of participants

SECONDARY OUTCOMES:
postoperative constipation | one year
  number of patients
postoperative uroschesis | one year
  number of patients
intestinal obstruction | one year
  number of patients
surgical wound infection | one year
  number of patients

OTHER OUTCOMES:
dyspareunia | one year
  number of patients

CONTACTS AND LOCATIONS:
Overall Officials: Yao Shuzhong, MD, Study Director — First Affiliated Hospital of Sun Yat-sen University